CLINICAL TRIAL: NCT01260077
Title: Steady State Vestibular Evoked Myogenic Potentials
Status: Completed | Type: Observational
Sponsor: Universidade Estadual de Ciências da Saúde de Alagoas (Other)
Responsible Party: PhD Pedro de Lemos Menezes, Professor, UNCISAL
Other Study IDs: CEP_UNCISAL_1010/2009
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2009-02

CONDITIONS: Normal Vestibular Evoked Potentials in Frequency Domain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Experimental group: The sample was composed of 78 individuals (156 ears), 40 females (80 ears) and 38 males (76 ears).

SUMMARY:
Objective: At present, vestibular evoked myogenic potentials are analyzed only in the time domain. A technique to evaluate this potential in the frequency domain could provide more information, but has only been applied within the last year. Design and Study Sample: In this study we recorded vestibular evoked myogenic potential in the time domain, in 156 ears of 78 normal-hearing young adults, at frequencies of 250, 500, 1000 and 2000 Hz, with intensity of 90 dB nHL. Next, the steady state vestibular evoked myogenic potential was recorded at the same carrying frequencies, modulated at 20, 37, 40, 43, 70, 77 and 80 Hz. Results: The responses found by modulated frequency, regardless of carrier, recorded a higher presence of peaks and mean amplitudes between 20 and 70 Hz, especially at 40 Hz. Conclusions: The results show that the observation technique in the frequency domain is feasible and shows a strong association with the time domain for recording vestibular evoked myogenic potentials, at carrying frequencies of 250, 500, 1000 or 2000 Hz.

ELIGIBILITY:
Inclusion criteria: age between 18 and 35 years and auditory threshold less than or equal to 20 dBHL, between 0.5 and 8 kHz, with inter-ear frequency difference less than or equal to 10 dB.

Exclusion criteria were: exposure to occupational or leisure noise; otological surgery; more than three ear infections within the last year; use of ototoxic medication; buzzing in the ear, vertigo, dizziness or other cochlear-vestibular symptoms ; presence of systemic alterations that could contribute to cochlear-vestibular pathologies, such as diabetes, hypertension, dyslipidemias and/or hormonal alterations.

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Normal subjects.
Sampling Method: Probability Sample

PRIMARY OUTCOMES:
A technique to evaluate vestibular evoked myogenic potential in the frequency domain

REFERENCES:
- [Derived] de Oliveira AC, Pereira LD, Colafemina JF, de Lemos Menezes P. Amplitude modulated vestibular evoked myogenic responses: a study of carrier and modulating frequencies. Acta Otolaryngol. 2014 Aug;134(8):796-801. doi: 10.3109/00016489.2014.909605. Epub 2014 Jun 9. PMID 24909625